CLINICAL TRIAL: NCT03184792
Title: Activity Dependent Rehabilitation Via Transcutaneous Electrical Spinal Stimulation to Restore Upper Extremity Functions in Spinal Cord Injury
Brief Title: Transcutaneous Electrical Spinal Stimulation to Restore Upper Extremity Functions in Spinal Cord Injury
Acronym: ADDRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Chet Moritz, Associate Professor, Rehabilitative Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002985
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury Cervical; Upper Extremity Dysfunction
Keywords: Spinal electrical stimulation
MeSH Terms: interventions — Physical Therapy Modalities; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups:
  Group 1.) Six weeks of "Physical therapy only" (Arm A) as the first intervention and then 6 weeks of "Transcutaneous spinal stimulation & Physical therapy" (Arm B) as the second intervention.
  Group 2.) Six weeks of "Transcutaneous spinal stimulation & Physical therapy" (Arm B) as the first intervention, and then "Physical therapy only" (Arm A) as the second intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Physical therapy only (Arm A) (Active Comparator): Physical therapy that targets the rehabilitation of upper extremity functions
  Interventions: Other: Physical therapy
- Transcutaneous cervical electrical stimulation combined with physical therapy (Arm B) (Experimental): Application of Transcutaneous cervical electrical stimulation combined with physical therapy that targets the rehabilitation of upper extremity functions
  Interventions: Device: Transcutaneous spinal stimulation; Other: Physical therapy

INTERVENTIONS:
Device: Transcutaneous spinal stimulation — Non-invasive electrical stimulation of cervical spinal cord over the skin
  Arms: Transcutaneous cervical electrical stimulation combined with physical therapy (Arm B)
Other: Physical therapy — Physical therapy to improve arm and hand functions
  Other Names: Exercise therapy

SUMMARY:
Stimulation of the spinal cord may induce the growth and reorganization of neural pathways leading to the re-animation of paralyzed limbs. Growing evidence indicates that electrical spinal cord stimulation improves motor functions immediately via modulating the excitability of spinal circuitry in patients with spinal cord injury. Recently, a novel, non-invasive, well-tolerated and painless transcutaneous electrical stimulation strategy was demonstrated to be effective for improving lower limb motor function in healthy individuals and in patients with spinal cord injury. The investigators hypothesize that transcutaneous cervical electrical stimulation can enhance conscious motor control and functions of hand and arm via neuromodulation of spinal network.

This study is a prospective efficacy trial of transcutaneous cervical electrical stimulation for improving upper limb function in patients with traumatic or degenerative cervical spinal cord injury. Transcutaneous electrical spinal stimulation device is not regulated by the United States Food and Drug Administration for treatment of spinal cord injury.

The interventions include either transcutaneous cervical spinal electrical stimulation combined with physical therapy or physical therapy only. The order of the interventions will be randomized for each subject in a delayed cross-over design. Total duration of the study is 6 months, including 4 weeks baseline measurements, 8 weeks intervention and 12 weeks follow-up. Both immediate and lasting improvements in hand motor and sensory function via transcutaneous cervical spinal stimulation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Cervical (C7 or higher) spinal cord injury at least 1-year duration
* Incomplete spinal cord injury (American Spinal Injury Association Impairment Scale (AIS) C or D)
* Between 21 and 70 years of age
* Difficulty with hand functions in activities of daily living (e.g. dressing, grooming, feeding)
* Stable medical condition without cardiopulmonary disease or frequent autonomic dysreflexia that would contraindicate participation in upper extremity rehabilitation or testing activities
* Capable of performing simple cued motor tasks
* Ability to attend 2 to 5 sessions of weekly physical therapy sessions and testing activities
* Adequate social support to be able to participate in weekly training and assessment sessions for the duration of 6 months within the study period.
* Ability to read and speak English

Exclusion Criteria:

* Autoimmune etiology of spinal cord dysfunction/injury
* History of additional neurologic disease, such as stroke, multiple sclerosis, traumatic brain injury, etc.
* Peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy, etc.)
* Rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
* Significant medical disease; including uncontrolled systemic hypertension with values above 170/100 mmHg; cardiac or pulmonary disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation.
* Active cancer
* Cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention
* Unhealed fracture, contracture, pressure sore, or urinary tract infection or other illnesses that might interfere with upper extremity rehabilitation or testing activities
* Any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician
* Pregnancy
* Tendon or nerve transfer surgery in the upper limbs
* Botulinum toxin injections in the prior 6 months
* Dependent on ventilation support
* Implanted stimulator (e.g. vagus nerve stimulator, pacemaker, cochlear implant, etc).
* Has depression or anxiety based on Patient Health Questionnaire and General Anxiety Disorder-7 item Questionnaire
* Diagnosed with syringomyelia
* Alcohol and/or drug abuse.
* Cognitive impairment based on Short Portable Mental Status Questionnaire
* Unable to read and/or comprehend the consent form.
* Unable to understand the instructions given as part of the study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chet T Moritz, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We use advertisement flyers and information sheets that will be clearly displayed in the neurosurgery and rehabilitation outpatient departments at the University of Washington, for all to see. Recruitment began on December 1, 2017, and concluded on December 1, 2023.
Groups:
- Group 1 (Cross-over Intervention arm sequence: AB): The sequence of cross-arm intervention for Group 1 will be as follows: "Physical therapy only (Arm A) first" and "Transcutaneous Spinal Cord Stimulation combined with Physical Therapy (Arm B) second."
- Group 2 (Cross-over Intervention arm sequence: BA): The sequence of cross-arm intervention for Group 2 will be as follows: "Transcutaneous Spinal Cord Stimulation combined with Physical Therapy (Arm B) first" and "Physical therapy only (Arm A) second."
Period: Overall Study
Arm/Group | Group 1 (Cross-over Intervention arm sequence: AB) | Group 2 (Cross-over Intervention arm sequence: BA)
Started | 7 (Group 1 (Cross-over intervention arm sequence AB): 7 participants received "Physical therapy only (Arm A)" as the FIRST intervention, and "Transcutaneous spinal stimulation & Physical therapy (Arm B)" as the SECOND intervention.) | 8 (Group 2 (Cross-over intervention arm sequence BA): 8 participants enrolled to receive "Transcutaneous spinal stimulation & Physical therapy (Arm B)" as the FIRST intervention, then Physical therapy only (Arm A)" as the SECOND intervention.)
Completed | 5 (In Group 1 (Cross-over intervention sequence is AB), 5 participants completed the study.) | 6 (In Group 2 (Cross-over intervention arm sequence is BA), 6 participants completed the study.)
Not Completed | 2 | 2
Not completed — Pandemic | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (Cross-over Intervention arm sequence: AB) - Active Comparator: The sequence of cross-arm intervention for Group 1 will be as follows: "Physical therapy only (Arm A) first" and "Transcutaneous Spinal Cord Stimulation combined with Physical Therapy (Arm B) second."
  Physical Therapy only is the active comparator intervention.
- Group 2 (Cross-over Intervention arm sequence: BA) - Experimental: The sequence of cross-arm intervention for Group 2 will be as follows: "Transcutaneous Spinal Cord Stimulation combined with Physical Therapy (Arm B) first" and "Physical therapy only (Arm A) second."
  Transcutaneous Spinal Cord Stimulation, combined with physical therapy, is the experimental intervention.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Cross-over Intervention arm sequence: AB) - Active Comparator | Group 2 (Cross-over Intervention arm sequence: BA) - Experimental | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14) | 60 (6) | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
International Standards for Neurological Classification of SCI (ISNCSCI) [Mean (Standard Deviation); unit: units on a scale] — International Standards for Neurological Classification of Spinal Cord Injury
  Subscale 1: Myotomal-based Motor Examination - measures the motor function of the extremities. The minimum score is zero, and the maximum score is 100. Higher scores represent better outcomes.
  Subscale 2: The Dermatomal-based Sensory Examination - measures the sensory function of the whole body dermatomes. The minimum score is zero, and the maximum score is 224. Higher scores represent better outcomes.
  units on a scale
    Subscale 1: Myotomal-based Motor Examination | 50.1 (21.5) | 49.8 (15.0) | 49.9 (17.8)
    Subscale 2:Dermatomal-based Sensory Examination | 111.0 (43.3) | 113.8 (36.4) | 112.4 (35.8)

OUTCOME MEASURES:

1. Primary Outcome: Graded and Redefined Assessment of Strength, Sensibility and Prehension Test (GRASSP Test)
Description: GRASSP is a clinical impairment measurement tool that quantifies hand impairment caused by cervical spinal cord injury. The tool measures three domains of function: strength (manual muscle strength testing), sensibility (Semmes-Weinstein monofilament sensation test), and prehension (ability and performance to generate various grasp and pinch movements using a water bottle, jar, key, pegs, coins, and nuts).
  The total score is calculated as the sum of the subscale scores. The minimum score is zero, and the maximum score is 232 points. Higher Scores mean a better outcome.
  Score change before and after each intervention is calculated.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score change before and after
Groups:
- Physical Therapy only: All participants, when they receive the "physical therapy only" intervention arm.
- Transcutaneous Spinal Cord Stimulation combined with Physical Therapy: All participants, when they receive Transcutaneous Spinal Cord Stimulation combined with Physical Therapy
Arm/Group | Physical Therapy only | Transcutaneous Spinal Cord Stimulation combined with Physical Therapy
Number analyzed (Participants) | 11 | 11
score change before and after | 4.5 (4.1) | 19.4 (6.3)
Statistical Analysis 1: Comparison: Physical Therapy only vs Transcutaneous Spinal Cord Stimulation combined with Physical Therapy; Test type: Superiority; p < 0.000, ANOVA; Mean Difference (Final Values) = 9.5, 95% CI 2-sided [6.6 to 12.4]
Statistical Analysis 2: Comparison: Physical Therapy only vs Transcutaneous Spinal Cord Stimulation combined with Physical Therapy; Test type: Superiority; p = 0.010, t-test, 2 sided; Median Difference (Final Values) = 10.4, 95% CI 2-sided [3.7 to 17.0]

2. Secondary Outcome: International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Examination
Description: International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Examination Subscale 1: Myotomal-based Motor Examination - measures the motor function of the extremities. The minimum score is zero, and the maximum score is 100. Higher scores represent better outcomes.
  Subscale 2: The Dermatomal-based Sensory Examination - measures the sensory function of the whole body dermatomes. The minimum score is zero, and the maximum score is 224. Higher scores represent better outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Transcutaneous Spinal Cord Stimulation combined with Physical Therapy: All participants, when they receive the "Transcutaneous Spinal Cord Stimulation combined with Physical Therapy" intervention arm.
Arm/Group | Physical Therapy only | Transcutaneous Spinal Cord Stimulation combined with Physical Therapy
Number analyzed (Participants) | 11 | 11
score on a scale
  Subscore 1: Myotomal-based Motor Examination | 0.5 (0.8) | 5.5 (2.3)
  Subscale 2: The Dermatomal-based Sensory Examination | 1.6 (5.2) | 6.4 (9.5)
Statistical Analysis 1: Comparison: Physical Therapy only vs Transcutaneous Spinal Cord Stimulation combined with Physical Therapy; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Grip and Pinch Strength
Description: Hand strength measurement by dynamometry.
  The change in strength (improvement) before and at the end of each intervention arm is calculated.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Physical therapy only | Transcutaneous Spinal Cord Stimulation combined with Physical Therapy
Number analyzed (Participants) | 11 | 11
kilogram | 3 (2) | 12 (4)

4. Secondary Outcome: Numeric Pain Rating Scale
Description: Patient reported pain rating on a 0 to 10 scale. The mean score change (improvement) before and at the end of each intervention arm is calculated.
  Zero means no pain, 10 means the worst pain one can imagine. Higher scores mean worse pain.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | physical therapy only | Transcutaneous Spinal Cord Stimulation combined with Physical Therapy
Number analyzed (Participants) | 11 | 11
score on a scale | 4.0 (1.1) | 2.0 (0.5)

5. Secondary Outcome: Penn Spasm Score
Description: Patient-reported spasm rating. Scores are mild (0), moderate (1), and severe (2).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Physical therapy only: All participants, while they receive "Physical Therapy only" intervention arm.
- Transcutaneous Spinal Cord Stimulation combined with Physical Therapy: All participants, while they receive "Transcutaneous Spinal Cord Stimulation combined with Physical Therapy" intervention arm.
Arm/Group | Physical therapy only | Transcutaneous Spinal Cord Stimulation combined with Physical Therapy
Number analyzed (Participants) | 11 | 11
score on a scale | 1.5 (0.5) | 1.0 (0)

6. Secondary Outcome: Spinal Cord Independence Measure (SCIM)
Description: Clinician-administered disability questionnaire for patients with spinal cord lesions.
  The total SCIM scores range from 0 to 100. Higher scores mean better outcomes. Score change (improvement) relative to baseline or previous intervention arm is calculated.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Physical therapy only: All participants, when they receive "Physical Therapy Only" intervention arm.
- ranscutaneous Spinal Cord Stimulation combined with Physical Therapy: All participants, when they receive the "Transcutaneous Spinal Cord Stimulation combined with Physical Therapy" intervention arm.
Arm/Group | Physical therapy only | ranscutaneous Spinal Cord Stimulation combined with Physical Therapy
Number analyzed (Participants) | 11 | 11
score on a scale | 0.2 (0.4) | 3.2 (2.2)

7. Secondary Outcome: World Health Organization-Quality of Life - (WHO-QoL-BREF)
Description: Patient-reported quality of life scale. A higher score indicates a higher quality of life. Score change (improvement) relative to baseline or prior intervention arm is calculated.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical therapy only | Transcutaneous Spinal Cord Stimulation combined with Physical Therapy
Number analyzed (Participants) | 11 | 11
score on a scale | 4.3 (7.7) | 12.5 (8.9)

ADVERSE EVENTS:
Time Frame: 6 years
Description: The intervention carries a low risk of mild adverse events. For that reason, serious adverse events were not expected.
Groups:
- Arm A: "Physical therapy only": Physical therapy: Physical therapy to improve arm and hand functions
- Arm B: "Transcutaneous spinal stimulation & Physical therapy": Transcutaneous spinal stimulation: Non-invasive electrical stimulation of the cervical spinal cord over the skin combined with Physical therapy to improve arm and hand functions.
Arm/Group | Arm A: "Physical therapy only" | Arm B: "Transcutaneous spinal stimulation & Physical therapy"
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT03184792/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT03184792/SAP_001.pdf